CLINICAL TRIAL: NCT00102050
Title: A Double-Blind, Randomized, Parallel Group, Placebo-Controlled Study to Evaluate the Safety and Efficacy of NM-702 in Subjects With Intermittent Claudication
Brief Title: Efficacy and Safety of NM-702 Tablets for the Treatment of Intermittent Claudication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nissan Chemical Industries (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-IC-0201
Record Dates: First submitted 2005-01-19; First posted 2005-01-20 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease
Keywords: NM-702 tablets; intermittent claudication; peripheral; arterial; vascular; peripheral arterial disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Peripheral Arterial Disease | interventions — 4-bromo-6-(3-(4-chlorophenyl)propoxy)-5-(3-pyridylmethylamino)-3(2H)-pyridazinone hydrochloride; Phosphodiesterase Inhibitors

INTERVENTIONS:
Drug: NM-702 (phosphodiesterase inhibitor)

SUMMARY:
NM-702 oral tablets are being developed for the treatment of Intermittent Claudication, a primary early stage indication of peripheral arterial disease (PAD). This trial is designed to assess the safety and efficacy of 4 mg and/or 8 mg NM-702 taken twice a day (BID) for 24 weeks to see if it improves peak walking time (PWT) more than placebo for the treatment of Intermittent Claudication.

DETAILED DESCRIPTION:
NM-702 oral tablets are being developed for the treatment of Intermittent Claudication, a primary early stage indication of peripheral arterial disease (PAD). This trial is designed to assess the safety and efficacy of 4 mg and/or 8 mg NM-702 BID for 24 weeks to see if it improves peak walking time (PWT) more than placebo for the treatment of Intermittent Claudication.

ELIGIBILITY:
Inclusion Criteria:

* Stable, symptomatic, intermittent claudication due to occlusive atherosclerotic disease of the lower extremities
* Median treadmill peak walking time between 90 and 600 seconds

Exclusion Criteria:

* Symptoms of limb threatening ischemia (ischemic rest pain, ischemic ulceration and/or gangrene)
* Clinically significant pulmonary, neurological or skeletal dysfunction (e.g., lumbar canal stenosis, emphysema, uncontrolled angina, multiple sclerosis, or gait altering amputation) that would directly interfere or limit exercise testing
* Subjects who have had, or will require, a peripheral revascularization procedure within 12 weeks prior to or following treatment initiation.
* A resting blood pressure greater than 150/100 and other clinically significant results.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2003-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Improvement in peak walking time at 24 weeks

SECONDARY OUTCOMES:
Improvement in claudication onset time at 24 weeks
Health status survey questionnaire
Walking impairment questionnaire

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Investigator, Long Beach, California
  - Investigator, Riverside, California
  - Investigator, San Diego, California
  - Investigator, San Francisco, California
  - Investigator, Torrance, California
  - Investigator, Clearwater, Florida
  - Investigator, Coral Gables, Florida
  - Investigator, Jacksonville, Florida
  - Investigator, Springfield, Illinois
  - Investigator, Shawnee Mission, Kansas
  - Investigator, New Orleans, Louisiana
  - Investigator, New York, New York
  - Investigator, Durham, North Carolina
  - Investigator, Toledo, Ohio
  - Investigator, Warwick, Rhode Island
  - Investigator, San Antonio, Texas
  - Investigator, Tacoma, Washington